CLINICAL TRIAL: NCT00674661
Title: Safety and Effectiveness of the UV-X System for Corneal Collagen Cross-Linking in Eyes With Corneal Ectasia After Refractive Surgery
Brief Title: Corneal Collagen Cross-Linking for Ectasia (CXL)
Acronym: CXL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UVX-003
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Ectasia
Keywords: ectasia; cross-linking; crosslinking; cornea; riboflavin; UVA
MeSH Terms: conditions — Dilatation, Pathologic; Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corneal Collagen Cross-linking (CXL) Treatment Group (Active Comparator): riboflavin ophthalmic solution and UVA irradiation
  Interventions: Drug: riboflavin ophthalmic solution; Device: UVA Irradiation
- Control Group (Sham Comparator): riboflavin opthalmic solution without UVA irradiation
  Interventions: Drug: riboflavin ophthalmic solution

INTERVENTIONS:
Drug: riboflavin ophthalmic solution — riboflavin 0.1% ophthalmic solution (approximately 32 drops, or 1.6 mL)
Device: UVA Irradiation — UVA light (365 nm at an irradiance of 3 mW/cm2) for 30 minutes
  Other Names: UV-X™ Illumination System
  Arms: Corneal Collagen Cross-linking (CXL) Treatment Group

SUMMARY:
Prospective, randomized multicenter study to determine the safety and effectiveness of performing corneal collagen cross-linking (CXL) using riboflavin and UVA light in eyes with ectasia after refractive surgery.

DETAILED DESCRIPTION:
Subjects are randomized to a control group or a treatment group, with the control group crossed over to the treatment group at the 3 month visit. Corneal collagen cross-linking is performed as a single treatment. Subjects are followed for 12 months after the procedure to evaluate the long term effects of corneal collagen cross-linking.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ectasia after refractive surgery
* Documented ectasia on Pentacam or topography map
* BSCVA worse than 20/20
* Must complete all study visits

Exclusion Criteria:

* History of delayed wound healing
* History of corneal melt or corneal dystrophy

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2007-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hersh, MD, Principal Investigator — Cornea and Laser Eye Institute
Locations (10):
- United States (10):
  - Shiley Eye Center, La Jolla, California
  - Gordon -Weiss Vision Institute, San Diego, California
  - Center for Excellence in Eye Care, Miami, Florida
  - Price Vision Group, Indianapolis, Indiana
  - Durrie Vision, Kansas City, Kansas
  - Wilmer Eye Institute at Johns Hopkins University, Baltimore, Maryland
  - Minnesota Eye Consultants, Minneapolis, Minnesota
  - Cornea & Laser Eye Institute; Hersh Vision Group, Teaneck, New Jersey
  - Edward Harkness Eye Institute at Columbia University Medical Center, New York, New York
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York

REFERENCES:
- [Derived] Greenstein SA, Fry KL, Hersh PS. Effect of topographic cone location on outcomes of corneal collagen cross-linking for keratoconus and corneal ectasia. J Refract Surg. 2012 Jun;28(6):397-405. doi: 10.3928/1081597X-20120518-02. PMID 22692521

RESULTS

PARTICIPANT FLOW:
Groups:
- Corneal Collagen Cross-linking (CXL) Treatment Group: riboflavin ophthalmic solution and UVA irradiation (365 nm at an irradiance of 3 mW/cm2) for 30 minutes
Period: Overall Study
Arm/Group | Corneal Collagen Cross-linking (CXL) Treatment Group | Control Group
Started | 67 | 63
Completed | 56 | 48
Not Completed | 11 | 15
Not completed — Other | 5 | 7
Not completed — Lost to Follow-up | 6 | 3
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corneal Collagen Cross-linking (CXL) Treatment Group | Control Group | Total
Number analyzed (Participants) | 67 | 63 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 63 | 130
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 16 | 39
  Male | 44 | 47 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 18 | 18 | 36
  Unknown or Not Reported | 40 | 36 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 50 | 45 | 95
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Maximum Keratometry (Kmax)
Description: The primary efficacy parameter was corneal curvature, as measured by maximum keratometry (Kmax) in the study eyes. Study success was defined as a difference of ≥1 D in the mean change in Kmax from baseline to 12 months between the CXL group and control group. Keratometry was measured manually and by pentacam.
Time Frame: baseline,12 months
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Corneal Collagen Cross-linking (CXL) Treatment Group | Control Group
Number analyzed (Participants) | 67 | 63
diopters | -0.5 (2.2) | 0.5 (2.3)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Corneal Collagen Cross-linking (CXL) Treatment Group | Control Group
Serious Adverse Events (participants affected / at risk) | 1/67 | 0/63
Other Adverse Events (participants affected / at risk) | 59/67 | 21/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corneal Collagen Cross-linking (CXL) Treatment Group (N=67) | Control Group (N=63)
Corneal epithelium defect (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corneal Collagen Cross-linking (CXL) Treatment Group (N=67) | Control Group (N=63)
Corneal opacity (Eye disorders) | 40 (45) | 1 (1)
Eye pain (Eye disorders) | 18 (19) | 0 (0)
Corneal epithelium defect (Eye disorders) | 14 (18) | 2 (2)
Punctate keratitis (Eye disorders) | 13 (13) | 2 (3)
Dry eye (Eye disorders) | 11 (12) | 3 (3)
Photophobia (Eye disorders) | 11 (12) | 0 (0)
Vision blurred (Eye disorders) | 11 (11) | 4 (4)
Eye irritation (Eye disorders) | 7 (7) | 0 (0)
Visual acuity reduced (Eye disorders) | 7 (7) | 1 (1)
Corneal striae (Eye disorders) | 5 (6) | 3 (3)
Lacrimation increased (Eye disorders) | 5 (5) | 0 (0)
Ocular discomfort (Eye disorders) | 5 (5) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 4 (4) | 3 (3)
Eyelid oedema (Eye disorders) | 4 (4) | 1 (1)
anterior chamber flare (Eye disorders) | 3 (3) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 3 (3) | 1 (1)
keratitis (Eye disorders) | 3 (3) | 0 (0)
Meibomian gland dyisfunction (Eye disorders) | 3 (4) | 2 (2)
Ocular hyperaemia (Eye disorders) | 3 (3) | 1 (1)
Visual impairment (Eye disorders) | 3 (3) | 1 (1)
Anterior chamber cell (Eye disorders) | 2 (2) | 0 (0)
Asthenopia (Eye disorders) | 2 (2) | 0 (0)
Corneal oedema (Eye disorders) | 2 (2) | 0 (0)
Glare (Eye disorders) | 2 (2) | 0 (0)
Halo vision (Eye disorders) | 2 (2) | 0 (0)
Corneal abrasion (Eye disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site has the right to publish or communicate study results upon the earlier of: (a) publication of a multi-center publication of the Study results coordinated by Sponsor; or (b) submission of the Study data by Sponsor to the FDA; provided that the Sponsor reviews the proposed communication of results within ninety (90) days in advance of its release. Sponsor can request delay of publication or data release to allow for filing of patent application prior to the publication or release.